CLINICAL TRIAL: NCT04462354
Title: Pancreatic Anastomosis After Duodenopancreatectomy: Pancreatogastrostomy Versus Blumgart Anastomosis: Prospective, Randomized and Multicentric Study
Brief Title: Pancreatic Anastomosis After Duodenopancreatectomy
Acronym: PANGASBLUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PANGASBLUM
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Anastomotic Leak; Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pancreatogastric anastomosis. (Active Comparator)
  Interventions: Procedure: Pancreatogastric anastomosis.
- Blumgart Anastomosis (Experimental)
  Interventions: Procedure: Blumgart Anastomosis

INTERVENTIONS:
Procedure: Blumgart Anastomosis — Patients undergoing cephalic duodenopancreatectomy, reconstructing pancreatic-enteric communication by Blumgart anastomosis
  Arms: Blumgart Anastomosis
Procedure: Pancreatogastric anastomosis. — Patients undergoing cephalic duodenopancreatectomy, reconstructing pancreatic-enteric communication by Pancreatogastric anastomosis.
  Arms: Pancreatogastric anastomosis.

SUMMARY:
A national, multicenter, randomized, prospective, parallel group clinical study to evaluate two therapeutic strategies (invaginating pancreatogastric anastomosis versus Blumgart anastomosis).

DETAILED DESCRIPTION:
Background: Postoperative pancreatic fistula is currently the most frequent complications after duodenopancreatectomy. There are currently no RCT comparing two of the most frequently used method of pancreato-enteric anastomosis (invaginating pancreatogastric anastomosis versus Blumgart anastomosis)

Hypothesis: in patients with resectable pancreatic and periampullary tumors, performing a Blumgart (AB) anastomosis for pancreatoenteric reconstruction after duodenopancreatectomy decreases the rate of postoperative pancreatic fistula (PPF) compared to to pancreatogastric anastomosis.

Main goal: To comparatively evaluate the rate of PPF in patients with pancreatic and periampullary tumors undergoing cephalic duodenopancreatectomy after reconstruction with Blumgart anastomosis or pancreatogastric anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Diagnosis of pancreatic and periampullary tumor pathology that requires pancreatoduodenectomy
* Signature of informed consent by the patient or his legal representative

Exclusion Criteria:

* Patients in whom liver metastases or peritoneal carcinomatosis are detected during surgery.
* Patients in whom tumor resection is ultimately not achieved due to intraoperative evidence that the tumor is locally advanced, unresectable.
* Patients with macroscopic residual tumor (R2).
* High risk patients with severe pathology (ASA IV) according to the American Association of Anesthetists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula rate (PPF) | 3 months
  The post-operative pancreatic fistula (PPF) rate will be measured using the definition of the International Study Group of Pancreatic Fistula (ISGPF) : any measurable amount of fluid from a drain placed during the operation or percutaneously, with an amylase concentration greater than three times the plasma value.

SECONDARY OUTCOMES:
Bleeding | 3 months
  According to the definition of the International Study Group on Pancreatic Surgery. which grades the severity of bleeding according to the clinical situation, diagnosis and need for treatment.
Gastric Emptying Delay (GED) | 3 months
  According to the definition of the International Study Group on Pancreatic Surgery, which establishes the existence of GED when a nasogastric tube is needed for more than 3 days or is placed from the third day of the postoperative period, as well as intolerance to an oral diet at the end of the first postoperative week.
Biliary Fistula | 3 months
  According to the definition of the International Study Group of Liver Surgery, which defines it as any measurable amount of fluid from a drain placed during the operation or percutaneously, with a concentration of bilirubin greater than three times the plasma value as of the third post-operative day.
Other complications. | 3 months
  All complications that may occur during the first 90 days of the postoperative period (including the mortality rate) should be collected and classified according to the Clavien-Dindo classification and the Comprehensive Complication Index (CCI)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain